CLINICAL TRIAL: NCT00869791
Title: A Study to Compare Pharmacokinetics and Pharmacodynamics of IPX066 to Standard Carbidopa-Levodopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IPX066-B08-11
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Other): Treatment Period 1:
  IPX066 - 7 days; Washout Period - 7 days;
  Treatment Period 2:
  IR CD-LD- 7 days
  Interventions: Drug: IPX066; Drug: IR CD-LD
- Sequence 2 (Other): Treatment Period 1:
  IR CD-LD - 7 days; Washout period - 7 days;
  Treatment Period 2:
  IPX066- 7 days
  Interventions: Drug: IPX066; Drug: IR CD-LD

INTERVENTIONS:
Drug: IPX066 — experimental drug product: extended-release carbidopa-levodopa capsules
  Other Names: ER CD-LD
Drug: IR CD-LD — active comparator: immediate-release carbidopa-levodopa capsules
  Other Names: immediate-release carbidopa-levodopa

SUMMARY:
This study evaluated the pharmacokinetics, motor effects, and assessed the safety of IPX066 compared with an immediate-release cabridopa-levodopa formulation in subjects with advanced Parkinson's disease.

DETAILED DESCRIPTION:
This was a randomized, multicenter, open-label, single and multiple oral dose, two-treatment, two-period, crossover study in LD-experienced subjects with Parkinson's disease (PD). Subjects received 7 days of one treatment (IPX066 or IR CD-LD) followed by an approximate 7-day washout period followed by another 7 days of the other treatment (IR CD-LD or IPX066). During the approximate 7-day washout period, subjects took their prestudy CD-LD regimen. Pharmacokinetic and efficacy/pharmacodynamic measurements were done on Days 1 and 8. Safety measures (electrocardiograms [ECGs], clinical laboratory tests, vital signs, adverse events [AEs], and concomitant medications) were evaluated over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female diagnosed with idiopathic PD, without any known cause for Parkinsonism.
2. If female and of childbearing potential, subject should be abstinent or continuing to practice and willing to continue throughout the study with appropriate contraceptives (defined as Nova ring, oral, injected, transdermal patch, implanted, or barrier). The subject must agree to take every precaution to ensure that pregnancy will not occur during the study.
3. At least 30 years old at the time of diagnosis of PD.
4. Mini Mental State Examination (MMSE) ≥ 26 at Screening Visit.
5. A responder to LD and currently being chronically treated with stable dosage of commercially available standard, orally disintegrating, or controlled-release CD LD for at least 1 month.
6. Must have predictable fluctuations between "on" and "off" states.
7. Hoehn and Yahr Stage I-IV when "on".
8. Able to provide informed consent and willing to sign Health Insurance Portability and Accountability Act (HIPAA) authorization.
9. Able and willing to comply with the protocol, including availability for all scheduled study visits and blood sample collections.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Diagnosed with atypical parkinsonism.
3. History, physical findings or laboratory results suggesting a diagnosis other than PD.
4. Allergic or nonresponsive to previous CD-LD therapy.
5. Any medical (e.g., liver or kidney impairment, peptic ulcer) or condition/history that, in the Investigator's opinion, may jeopardize the subject's safety.
6. Exposure to any investigational agent within 30 days prior to Visit 1.
7. Donated blood or plasma within 28 days.
8. Had prior functional neurosurgical treatment for PD (ablation or Deep Brain Stimulation).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (1):
- IMPAX Laboratories, Hayward, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser RA, Ellenbogen AL, Metman LV, Hsu A, O'Connell MJ, Modi NB, Yao HM, Kell SH, Gupta SK. Crossover comparison of IPX066 and a standard levodopa formulation in advanced Parkinson's disease. Mov Disord. 2011 Oct;26(12):2246-52. doi: 10.1002/mds.23861. Epub 2011 Jul 13. PMID 21755537
- See also: PebMed Abstract — http://www.ncbi.nlm.nih.gov/pubmed/21755537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects were screened. 8 were screen failures (did to not meet inclusion/exclusion criteria) and 27 were randomized. Date of first patient enrolled: November 25, 2008 Date last patient completed: June 11, 2009 The study was conducted at 6 sites in the United States.
Pre-assignment Details: 27 participants were enrolled, treated and completed the treatment with this protocol.
Groups:
- IPX066 First (7 Days), Washout (7 Days) Then IR CD-LD (7 Days): In this arm there were 2 treatment periods of one week each. During period 1, 14 subjects received 7 days of IPX066 first. Then subjects returned to their pre-study regimen during the washout period of approximately 1 week. This was followed by Period 2. During period 2, the 14 subjects received IR CD-LD for 7 days.
- IR CD-LD First ( 7 Days), Washout (7 Days) Then IPX066 (7days): In this arm there were 2 treatment periods of one week each. During period 1, 13 subjects received 7 days of IR CD-LD first. Then subjects returned to their pre-study regimen during the washout period of approximately 1 week. This was followed by Period 2. During period 2, the 13 subjects received IPX066 for 7 days.
Period: Period 1 Treatment for 7 Days
Arm/Group | IPX066 First (7 Days), Washout (7 Days) Then IR CD-LD (7 Days) | IR CD-LD First ( 7 Days), Washout (7 Days) Then IPX066 (7days)
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Period 2 Treatment for 7 Days
Arm/Group | IPX066 First (7 Days), Washout (7 Days) Then IR CD-LD (7 Days) | IR CD-LD First ( 7 Days), Washout (7 Days) Then IPX066 (7days)
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either IPX066 or IR CD-LD
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Measurements to Determine Cmax for Carbidopa (CD) and Levodopa (LD) Plasma Concentrations From Samples Collected Pre-dose and at Different Time Points on Day 1 and Day 8 of Periods 1 and 2 of Both Treatment Arms.
Description: For both treatment arms: Sequence 1 (IPX066, Washout, then IR CD-LD) and Sequence 2 (IR CD-LD, Washout, IPX066), blood samples for measurement of LD and CD plasma concentrations were collected pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, and 8 hours after dosing on Day 1 (referred to as Single-Dose data); and at pre-dose, 0.5, 1,1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing on Day 8 (referred to as Multiple-Dose data). Maximum (peak) drug concentration (Cmax in nanograms/milliliter) was estimated using Single-Dose data and Multiple-Dose data.
Time Frame: Day 1 and on Day 8 after a week of intervention in each treatment arm: Arm 1 (IPX066 first, washout, then CD-LD IR) and Arm 2 (CD-LD IR first, washout, then IPX066)
Population: The study was designed to assess the single and multiple-dose PK and PD of IPX066 and IR CD-LD in subjects with advanced PD.14 subjects first received IPX066 (Period 1), then IR CD-LD (Period 2). 13 Subjects first received IR CD-LD (Period 1), then IPX066 (Period 2). All 27 subjects that were treated in the study were included in the PK analyses.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Groups:
- IPX066: All participants who received IPX066 in either study period
- IR CD-LD: All participants who received IR CD-LD in either study period
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
nanogram/milliliter
  CD Cmax, Single-Dose | 238.852 (91.004) | 146.848 (58.787)
  CD Cmax, Multiple-Dose | 313.222 (167.924) | 167.515 (51.204)
  LD Cmax, Single-Dose | 3000.000 (1301.608) | 2356.444 (1080.541)
  LD Cmax, Multiple-Dose | 3807.037 (1547.120) | 2761.852 (1002.984)

2. Primary Outcome: Pharmacokinetics Measurements to Determine Tmax for Levodopa and Carbidopa Plasma Concentrations From Samples Collected Pre-dose and at Different Time Points on Day 1 and Day 8 of Periods 1 and 2 of Both Treatment Arms.
Description: For both treatment arms: Sequence 1 (IPX066, Washout, then IR CD-LD) and Sequence 2 (IR CD-LD, Washout, IPX066), blood samples for measurement of LD and CD plasma concentrations were collected pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, and 8 hours after dosing on Day 1 (referred to as Single-Dose data); and at pre-dose, 0.5, 1,1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing on Day 8 (referred to as Multiple-Dose data). Time of maximum drug concentration (Tmax in hours) was estimated using Single-Dose data and Multiple-Dose data.
Time Frame: Day 1 and on Day 8 after a week of intervention in each treatment arm: Arm 1 (IPX066 first, washout, then CD-LD IR) and Arm2 (CD-LD IR first, washout, then IPX066
Population: The study was designed to assess the single and multiple-dose PK and PD of IPX066 and IR CD-LD in subjects with advanced PD. 14 subjects first received IPX066 (Period 1), then IR CD-LD (Period 2). 13 Subjects first received IR CD-LD (Period 1), then IPX066 (Period 2). All 27 subjects that were treated in the study were included in the PK analyses.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
Hours
  CD Tmax Single-Dose | 2.944 (0.5604) | 2.296 (0.6086)
  CD Tmax Multiple-Dose | 3.815 (2.6390) | 5.685 (3.5711)
  LD Tmax Single-Dose | 2.037 (1.0735) | 0.870 (0.4921)
  LD Tmax Multiple-Dose | 4.407 (3.7597) | 3.611 (4.2161)

3. Primary Outcome: Pharmacokinetics Measurements to Determine Area Under the Concentration-time Curve for the Dosing Interval for LD and CD Concentrations From Blood Collected Pre-dose and at Different Time Points on Day 1 and Day 8 of Periods 1 and 2 of Treatment Arms.
Description: For both treatment arms: Sequence 1 (IPX066, Washout, then IR CD-LD) and Sequence 2 (IR CD-LD, Washout, IPX066), blood samples for measurement of LD and CD plasma concentrations were collected pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, and 8 hours after dosing on Day 1 (referred to as Single-Dose data); and at pre-dose, 0.5, 1,1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing on Day 8 (referred to as Multiple-Dose data). Area under the concentration-time curve for the dosing interval (AUC Tau) in hour*nanogram/milliliter was estimated using Single-Dose data and Multiple-Dose data.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
hour*nanogram/milliliter
  CD AUC Tau, Single-Dose | 917.067 (373.9147) | 401.694 (177.8239)
  CD AUC Tau, Multiple-Dose | 1344.436 (818.1622) | 449.584 (273.8498)
  LD AUC Tau, Single-Dose | 10902.194 (4619.2284) | 3881.298 (1586.9059)
  LD AUC Tau, Multiple-Dose | 13903.380 (6990.0405) | 4167.151 (1799.2567)

4. Secondary Outcome: 8-Hour Efficacy Using Day 1 Tapping
Description: Improvement in "Tapping: has been used as a surrogate endpoint for assessing subject being "On". Finger Tapping: the number of times the subject could tap two counter keys 20 cm apart alternately in 1 minute with the most affected arm assessed every 30 minutes on Day 1. Subjects performed the 60-second tapping measurement three times prior to dosing in the clinic, and at half-hour intervals through the 8-hour measurement period on Day 1 of each treatment period. More hours "On" during treatment represented better outcome. For the Tapping measurement, the protocol defined a 20% change from the average of the predose measurements as the time to "On." Each half-hour interval counted as 0.5 hour. Any measurement below a 20% improvement was considered time "Not On." If patient required redosing then primary analyses adjusted for redosing in calculating the results.
Time Frame: Day 1 of each treatment period - three times prior to dosing in the clinic, and at half-hour intervals through the 8-hour measurement period
Population: Analysis of covariance was the primary analysis conducted on the mean total Taps across the 8-hour measurement period, with the average of the three predose Tapping measurement values as a covariate.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
Hours | 4.74 (2.843) | 2.98 (2.436)

5. Secondary Outcome: 8-Hour Efficacy Using Day 1 Unified Parkinson's Disease Rating Scale Part III Score
Description: To determine efficacy on Day 1 the UPDRS (unified Parkinson's disease rating) Part III score, a clinician-scored measure of motor function, was collected immediately predose and 1, 2, 3, 4, 5, 6, 7 and 8 h post dose. The UPDRS Part III motor exam analyzes multiple motor functions like speech, facial expression, tremor, rigidity, movement, posture, gait etc. Each parameter is assigned values from 0 to 4, with 0 being normal and 4 being the most affected. The total range is 0 - 108, with lower scores indicating a better outcome.The average of post dose was calculated for day 1.
Time Frame: Pre dosing and at hourly intervals through the 8-hour measurement period on day 1
Population: Analysis of covariance was the primary analysis conducted on the mean UPDRS Part III across the 8-hour measurement period, with the predose UPDRS Part III value as a covariate. This analysis was repeated at each timepoint for completeness.
Measure: Mean (Standard Deviation); unit: UPDRS Part III Motor Score
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
UPDRS Part III Motor Score | 21.6 (9.81) | 25.5 (9.54)

6. Secondary Outcome: Result Summary of Day 1 Dyskinesia Evaluated by Investigator Assessment for Each Treatment Period
Description: To determine 8h efficacy on Day 1 the on site investigator assessments of "ON", "OFF" and "state of dyskinesia" for each subject was collected predose (-1, -0.5, and 0 hours) every 30 min for up to 8 hours after dosing . For all subjects duration of (1) OFF time (2) ON time without dyskinesia, (3) ON time with non-troublesome dyskinesia and (4) ON time with troublesome dyskinesia was calculated for both treatments. Definition of "ON" was based on a 20% change from predose measure, and the results were analyzed in the standard manner of a two way crossover design. The trial inclusion criteria included ability of subject to differentiate "ON" state from "OFF" state per investigator's assessment.
Time Frame: Predose and then every 30 min upto 8 h after dosing on Day of 1 of each treatment period
Population: For determining motor assessment of dyskinesia evaluated by investigator assessment a mixed-effect model was used with treatment, sequence, and period as factors and subjects within sequence as error term. The primary analysis was performed on the average of all times collected half hourly. Data for two patients was not collected, N25 instead of 27
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 25 | 25
Hours
  OFF time | 1.90 (1.588) | 4.44 (1.364)
  ON time without dyskinesia | 2.94 (2.468) | 2.36 (1.840)
  ON time with non-troublesome dyskinesia | 2.62 (2.242) | 0.90 (0.968)
  ON time with troublesome dyskinesia | 0.54 (1.070) | 0.28 (0.830)

7. Secondary Outcome: "Off" Time Hours Reported by Subjects Using Parkinson's Patient Diary
Description: Subjects recorded state of "OFF" time using the Parkinson's Patient Diary
Time Frame: Last 3 days of each treatment period, every 30 minutes over a 24-hour day beginning at 6:00 AM
Population: All treated patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IPX066 | IR CD-LD
Number analyzed (Participants) | 27 | 27
hours | 3.83 (2.80) | 5.83 (2.92)

ADVERSE EVENTS:
Time Frame: At each of the 4 study visits and follow-up with the subject by phone within 1 week of study exit.
Description: Safety measures (electrocardiograms [ECGs], clinical laboratory tests, vital signs, adverse events [AEs], and concomitant medications) were evaluated over the course of the study. The Investigators were specified in the protocol to follow each AE until resolution or stabilization and in accordance with Good Clinical Practice (GCP). Follow-up on these AEs were be recorded on the source documents and reported to IMPAX.
Groups:
- CD-LD IR: All participants who received IR CD-LD in either study period
Arm/Group | IPX066 | CD-LD IR
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/27 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPX066 (N=27) | CD-LD IR (N=27)
Sleepy (Nervous system disorders) | 1 (1) | 0 (0)
Choreiform Movements (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Feeling of Warth in Abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache - Frontal (Nervous system disorders) | 1 (1) | 0 (0)
Common Cold (Infections and infestations) | 0 (0) | 1 (1)
Dizziness after Taking Medication (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study include its relatively small size, multiple statistical testing, short study durations, and open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No